CLINICAL TRIAL: NCT03250767
Title: A Post-Market, Prospective, Multi-Center, Open-Label, Single Arm Clinical Evaluation of the Integra® Titan™ Modular Shoulder System Generation 2.5 for Primary Shoulder Joint Replacement
Brief Title: Clinical Evaluation of the Integra® Titan™ Modular Shoulder System Generation 2.5 for Primary Shoulder Joint Replacement
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not due to adverse events, complications, or device issues.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: T-TSS-003
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Osteo Arthritis Shoulders; Traumatic Arthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Integra Titan Modular Shoulder System 2.5
  Interventions: Device: Integra Titan Modular Shoulder System 2.5

INTERVENTIONS:
Device: Integra Titan Modular Shoulder System 2.5 — Primary Shoulder Joint Replacement

SUMMARY:
A post market, prospective, non-randomized, multi-center, open-label, clinical study using survivorship as the reference performance goal to study the safety and efficacy of the Titan Modular Shoulder System 2.5 when used for primary shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* For total shoulder arthroplasty, subjects must meet a, b, or c below:

  1. Severely painful and/or disabled joint resulting from osteoarthritis, traumatic arthritis or rheumatoid arthritis
  2. Fracture-dislocations of the proximal humerus where the articular surface is severely comminuted, separated from its blood supply or where the surgeon's experience indicates that alternative methods of treatment are unsatisfactory
  3. Other difficult clinical problems where shoulder arthrodesis or resection arthroplasty are not acceptable (e.g. -revision of a failed primary component)
* For shoulder hemiarthroplasty, subjects must meet any of the sub-criteria a - g below:

  1. Severely painful and/or disabled joint resulting from osteoarthritis, traumatic arthritis or rheumatoid arthritis
  2. Fracture-dislocations of the proximal humerus where the articular surface is severely comminuted, separated from its blood supply or where the surgeon's experience indicates that alternative methods of treatment are unsatisfactory
  3. Other difficult clinical problems where shoulder arthrodesis or resection arthroplasty are not acceptable (e.g. -revision of a failed primary component)
  4. Ununited humeral head fractures
  5. Avascular necrosis of the humeral head
  6. Rotator cuff arthropathy
  7. Deformity and/or limited motion

Exclusion Criteria:

* Absent, irreparable or nonfunctional rotator cuff or other essential muscles.
* Have an active local or systemic infection.
* Have inadequate bone stock in the proximal humerus or glenoid fossa for supporting the components.
* Have poor bone quality such as osteoporosis where there could be considerable migration of the prosthesis and/or a chance of fracture of the humerus or glenoid.
* Have a muscular, neurologic, or vascular deficiencies that compromise the affected extremity.
* Have a known sensitivity or allergic reaction to one or more of the implanted materials.
* Have a condition that may impair proper wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with shoulder arthritis requiring primary shoulder joint replacement
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Implant Survivorship | 2 years
  Implant survivorship defined as absence of device removal or revision

SECONDARY OUTCOMES:
Implant Survivorship | 1,5 and 10 years
  Implant survivorship defined as absence of device removal or revision
Relative change of Range of Motion (ROM) compared to baseline | up to 10 years
  Relative change of ROM compared to baseline
Relative change of Constant-Murley Score (CMS) compared to baseline | up to 10 years
  Relative change of CMS compared to baseline
Relative change of American Shoulder & Elbow Surgeons Score (ASES) compared to baseline | up to 10 years
  Relative change of ASES compared to baseline
Relative change of Single Assessment Numeric Evaluation (SANE) compared to baseline | up to 10 years
  Relative change of SANE compared to baseline
Relative change of Simple Shoulder Test (SST) compared to baseline | up to 10 years
  Relative change of SST compared to baseline
Relative change of Pain compared to baseline | up to 10 years
  Relative change of Visual Analogue Scale (VAS) Pain compared to baseline

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - John Hopkins University, Columbia, Maryland
  - Mississipi Bone and Joint Clinic, Starkville, Mississippi
  - The Research Foundation for The State University of New York (SUNY), Syracuse, New York
  - Westphal Orthopaedics, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Rothman Institute, Philadelphia, Pennsylvania